CLINICAL TRIAL: NCT00331565
Title: Investigations on the Influence of Bariatric Surgery on the Metabolism and Absorption of Atorvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ATORVA-06
Record Dates: First submitted 2006-05-29; First posted 2006-05-31 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery; Bioavailability; Bioequivalence; Atorvastatin; CYP's; P-gp; OATP
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

ARMS (1):
- Surgery (Experimental): Bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Gastric bypass, duodenal switch and sleeve surgery

SUMMARY:
Altered bioavailability of drugs will potentially affect both drug efficacy as well as safety. In patients subjected to bariatric surgery due to morbid obesity the gastro intestinal tract is considerably reconstructed and a change in drug bioavailability is very likely. Getting further knowledge on important mechanisms responsible for altered bioavailability would help in predicting clinically relevant consequences on different drugs.

In the present study we aim to investigate the effect of bariatric surgery on atorvastatin bioavailability. Atorvastatin is subjected to both extensive metabolism and drug transport and will potentially be a good predictor for mechanisms relevant for other drugs as well.

In addition will the expression of different enzymes and transporters be measured in the gastrointestinal tract and in the liver to elucidate on mechanism behind the eventual effects.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the effect of gastric bypass and BPD+DS operations on atorvastatin bioavailability.

Secondary objectives are to determine the relative change in atorvastatin bioavailability following gastric bypass as well as BPD+DS operations. In addition will the individual CYP3A4, CYP3A5 and P-gp activity in the different organs from where biopsies can be obtained be descriptively compared with atorvastatin pharmacokinetic variables.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for bariatric surgery.
* 18 years of age or older.
* Ongoing treatment with statin.
* Able and willing to donate GI-tract and liver biopsies.
* Signed informed consent.

Exclusion Criteria:

* Concomitant treatment with drugs and/or other factors that may influence atorvastatin pharmacokinetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
ratio of atorvastatin AUC0-8 between groups | june 2009

SECONDARY OUTCOMES:
Change in bioavailability of atorvastatin within each surgical technique will be analyzed as ratio of AUC0-8 from before to after surgery in accordance to the bioequivalence criteria of 80-125%. | june 2009
Descriptive comparison of mRNA expression of CYP3A4, CYP3A5, P-gp and OATP1B1 in different biopsies and atorvastatin and metabolites pharmacokinetics. | june 2009
Descriptive comparison of protein expression of CYP3A4, CYP3A5 and P-gp in different biopsies and atorvastatin and its metabolites pharmacokinetics. | december 2009
Descriptive listing of atorvastatin and metabolites concentrations in patients with different genotypes analyzed. It is anticipated that an exploratory analysis will be performed to compare the groups. | june 2009
Descriptive listing of the relationship between plasma and skeletal muscle as well as adipose tissue concentrations of atorvastatin and metabolites. | december 2009
Adverse events and serious adverse events will be listed. | june 2009

CONTACTS AND LOCATIONS:
Overall Officials: Rune Sandbu, MD, PhD, Principal Investigator — Hospital in Vestfold
Locations (1):
- Hospital in Vestfold, Tønsberg, Norway